CLINICAL TRIAL: NCT02030392
Title: "Stop the Pain"-A Multicenter, Randomized-controlled Study of a Cognitive-behavioral Intervention for Children With Functional Abdominal Pain
Brief Title: A Randomized-controlled Study of a Cognitive-behavioral Intervention for Children With Functional Abdominal Pain
Acronym: Stop-FAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Potsdam (Other)
Responsible Party: Principal Investigator, Petra Warschburger, Prof. Dr., University of Potsdam
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: WA1143/9-1; DRKS00005038 (Registry Identifier: DRKS)
Record Dates: First submitted 2013-10-28; First posted 2014-01-08 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Functional Abdominal Pain Syndrome; Abdominal Pain
Keywords: Functional abdominal pain; psychological intervention; quality of life; Randomized controlled trial; children
MeSH Terms: conditions — Abdominal Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention group (Experimental): IG participation in the cognitive-behavioral program "Stop the pain with Happy Pingu". The program compromises six weekly sessions for the children in small groups (90 min each) and 2 sessions for the parents (90 min each).
  Interventions: Behavioral: Intervention group
- Active control group (Active Comparator): CG participation in an information and education control group (physical well-being, health and gastrointestinal tract). The program of the control group compromises six weekly sessions for the children in small groups (90 min each) and 2 sessions for the parents (90 min each).
  Interventions: Behavioral: Active control group

INTERVENTIONS:
Behavioral: Intervention group — Cognitive-behavioral intervention
  Other Names: Stop the pain with Happy Pingu
  Arms: Intervention group
Behavioral: Active control group — Education and information
  Arms: Active control group

SUMMARY:
This trial aims to compare two training programs for children suffering functional abdominal pain. These two programs are comparable in number of sessions and group sizes, but show differences in content (very focused on pain management vs. more general information and support). Focus of the trial is the evaluation of "Stop the pain", which has shown high effectiveness in one first trial. This time, five clinics, experienced in diagnosis and treatment of childhood chronic abdominal pain, will take part. Children aged 7-12 years are eligible. The programs imply six weekly group sessions for the children and 2 parent evenings. The study group assumes that participation in "Stop the pain" will reduce pain experience and will improve the children's quality of life and coping strategies - up to 12 months after training.

DETAILED DESCRIPTION:
The trial aims to assess the efficacy of a cognitive-behavioral self-management program (intervention group, IG) compared to an equally extensive information-only control group (CG). The interventions contain 6 weekly group sessions and 2 parent meetings according to the cognitive-behavioral, manualized program "Stop the pain with Happy Pingu". Follow up per patient: 3- and 12 months. Children aged 7-12 years suffering functional abdominal pain (according to Rome III criteria H2a, H2b, H2d, H2d1) are eligible. Our primary hypothesis is that for patients in the IG the frequency and intensity of pain will be reduced more successfully and more sustainable than for children in the CG. Secondary hypotheses state that the IG will experience a higher increase in quality of life and psychosocial well-being compared to the active CG.

ELIGIBILITY:
Inclusion criteria for medical screening:

* aged 7-12 years
* abdominal pain for at least 2 months
* abdominal pain at least once per week
* unclear cause for abdominal pain

exclusion criteria for medical screening:

* very limited German language skills
* mental retardation
* adjuvant psychological treatment at point of medical screening
* participation in a trainingsprogram for abdominal pain in the 6 months prior to medical screening
* participation in a clinical trial which possibly may have effects on abdominal pain in the 4 weeks prior to medical screening
* at point of medical screening: therapy or medication for abdominal pain
* presentation of sibling aged 7-12 years

Inclusion Criteria for study participation:

* pain-predominant functional gastrointestinal disorders according to Rome-III
* criteria (H2a, H2b, H2d, H2d1)
* informed consent for study particiaption
* informed consent for audiotaping of trainings sessions
* no time constraints for participation in training groups

Exclusion Criteria for study participation:

* psychiatric disorder (internalizing) with primary treatment indication
* severe externalizing disorder

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 127 (Actual)
Dates: Start 2014-03-31 (Actual); Primary Completion 2017-07-07 (Actual); Study Completion 2017-07-07 (Actual)

PRIMARY OUTCOMES:
Change in Pain Symptoms | up to 21 days pre intervention, up to 21 days post intervention, 3 month-follow-up, 12 month-follow-up
  Primary efficacy endpoint is the frequency and intensity of pain (composite score) over the course of treatment and follow-up (pre, post, 3 and 12 months follow-up). This primary outcome will be assessed by pain diary in children's self-report (over 2 weeks).Statistically, the primary endpoint of the study is defined as the change of the logarithm of the area under the pain-intensity curve over one week from start of treatment to 12 month follow-up. The area under the pain intensity curve (auc) is a measure that reflects pain intensity as well as pain duration and pain frequency and thus can be understood as a composite measure of pain.

SECONDARY OUTCOMES:
Pain-related impairment | up to 21 days pre intervention, up to 21 days post intervention, 3 month-follow-up, 12 month-follow-up
  A measure for child's functional disability due to pain. The measure is one scale score and covers the level of impairment in everyday activitites due to abdominal pain by 12 items, e.g. reading, meeting friends, family life. The secondary outcome variable will be assessed by self-report questionnaire (pre, post, 3- and 12 months follow-up).
Health-related quality of life | up to 21 days pre intervention, up to 21 days post intervention, 3 month-follow-up, 12 month-follow-up
  The secondary outcome variable will be assessed by self-report questionnaire (pre, post, 3- and 12 months follow-up).
Pain-related coping and cognitions | up to 21 days pre intervention, up to 21 days post intervention, 3 month-follow-up, 12 month-follow-up
  The secondary outcome variable will be assessed by self-report questionnaire (pre, post, 3- and 12 months follow-up).

CONTACTS AND LOCATIONS:
Overall Officials: Petra Warschburger, Professor, Principal Investigator — University of Potsdam, Counselling Psychology
Locations (6):
- Germany (6):
  - University Medical Center, Pediatric Gastroenterology, Berlin
  - Children's Hospital "Prinzessin Margaret", Pediatric Gastroenterology, Darmstadt
  - University Medical Center, Pediatric Gastroenterology, Düsseldorf
  - Catholic Children's Hospital Hamburg Wilhelmstift, Hamburg
  - St. Vincenz Hospital, Paderborn
  - University Medical Center, Pediatric Gastroenterology, Ulm

REFERENCES:
- [Background] Gross M, Warschburger P. Evaluation of a cognitive-behavioral pain management program for children with chronic abdominal pain: a randomized controlled study. Int J Behav Med. 2013 Sep;20(3):434-43. doi: 10.1007/s12529-012-9228-3. PMID 22328460
- [Background] Groß, M. & Warschburger, P. (2013). Chronische Bauchschmerzen: Psychosoziale Belastung und behandlungsinduzierte Veränderungen in der Krankheitsbewältigung. Verhaltenstherapie, 23, 80-89. doi: 10.1159/000351215.
- [Background] Warschburger, P. & Groß, M. (2008). "Stopp den Schmerz" - ein kognitiv-behaviorales Behandlungsprogramm für Kinder mit Bauchschmerzen. Verhaltenstherapie, 18, 162-167.
- [Background] Warschburger P, Calvano C, Becker S, Friedt M, Hudert C, Posovszky C, Schier M, Wegscheider K. Stop the pain: study protocol for a randomized-controlled trial. Trials. 2014 Sep 11;15:357. doi: 10.1186/1745-6215-15-357. PMID 25212457
- [Derived] Warschburger P, Calvano C, Becker S, Ebinger F, Hudert C, Iven E, Posovszky C, Winter SM, Daubmann A, Ozga AK, Wegscheider K. Do Children With Functional Abdominal Pain Benefit More From a Pain-Specific Cognitive-Behavioral Intervention Than From an Unspecific Attention Control Intervention? Results of a Randomized Controlled Trial. Am J Gastroenterol. 2021 Jun 1;116(6):1322-1335. doi: 10.14309/ajg.0000000000001191. PMID 33767111
- See also: Homepage Counseling Psychology, Prof. Warschburger — http://www.psych.uni-potsdam.de/counseling/index-e.html
- See also: Description of research project — http://www.psych.uni-potsdam.de/counseling/research/fap-e.html